CLINICAL TRIAL: NCT05579847
Title: The Feasibility of an Educational and Monitoring Smart-Phone Application for Patients With Advanced Renal Cell Carcinoma Undergoing Combination Immunotherapy
Brief Title: Feasibility of a Smart-Phone App for Patients With Advanced Renal Cell Carcinoma Undergoing Combination Immunotherapy
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: MCC-21569
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Renal Cell Carcinoma Stage IV
Keywords: Kidney cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Participants: Participants with Stage IV Renal Cell Carcinoma will be recruited in the genitourinary medical oncology clinic at Moffitt Cancer Center. Upon consenting, participants will be provided with an mHealth interactive smart phone application.
  Interventions: Other: mHealth Smart Phone Application; Behavioral: eHEALS digital literacy test; Behavioral: Weekly Quiz; Behavioral: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire; Behavioral: Patient Post Intervention Survey

INTERVENTIONS:
Other: mHealth Smart Phone Application — The mHealth interactive application consists of educational intervention geared towards eligible patients who are receiving Nivolumab/ Pembro with Axitinib/Cabozantinib/Lenvatinib. These patients commonly experience immune-related side effects, higher rate of fatigue, high blood pressure, and palmar-plantar erythrodysesthesia. The educational intervention will consist of multiple modules covering relevant information on treatment and adverse events and provided over a six-week period through an mHealth platform. This educational intervention includes a patient-friendly algorithm for early detection and management of the most common adverse events in patients with advanced renal cell carcinoma receiving combination immunotherapy.
Behavioral: eHEALS digital literacy test — The eHEALS digital literacy test is an 8-item measure of eHealth literacy developed to measure the participants combined knowledge, comfort and perceived skills at finding, evaluating and applying electronic health information to health problems. The test is measured with a 5-point Likert scale with response options ranging from "strongly disagree" to "strongly agree." Total scores of the eHEALS are summed to range from 8 to 40, with higher scores representing higher self-perceived eHealth literacy.
Behavioral: Weekly Quiz — Participants will take a weekly true/false quiz to assess knowledge of their diagnosis, expected outcome and treatment associated adverse effects at baseline and longitudinally. Each quiz will be administered at the beginning of the week before the weekly educational content is available, then the same quiz will be administered after the educational content is reviewed by the patient. Each quiz will be scored based on the number of correct answers.
Behavioral: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire — The European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C-30) comprises 30 single questions, 24 of which are aggregated into nine multi-item scales, that is, five functioning scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. The remaining six single-item (dyspnea, appetite loss, sleep disturbance, constipation, diarrhea and the financial impact) scales assess symptoms. No item occurs in more than one scale.
  Scoring of the QLQ-C30 is performed according to QLQ-C30 Scoring manual. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient).
Behavioral: Patient Post Intervention Survey — The Patient Post Intervention Survey is a 7 question survey to help determine the effectiveness of the mHealth app. 3 questions are open fields for patient feedback, and 4 questions ask how often the app was used, how often the educational module was used and if the patient found it useful.

SUMMARY:
The purpose of the study is to test and understand acceptability and preliminary effectiveness of a mobile educational app specifically customized to patients with advanced Renal Cell Carcinoma (RCC) receiving therapy with combination immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stage IV Renal Cell Carcinoma
* Within 3 weeks from starting combination immune checkpoint blockade with tyrosine kinase inhibitor or multikinase inhibitor
* Estimated survival of 6 months or more
* Able to read and speak English

Exclusion Criteria:

* Unable to read or speak English
* Enrolled in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the genitourinary medical oncology clinic at Moffitt Cancer Center with Stage IV Renal Cell Carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2024-01-07 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Acceptability of Smart Phone Application | at 6 months
  Patient's acceptability of the smart phone application for education will be captured in the patient post education survey.

SECONDARY OUTCOMES:
Efficacy of Smart Phone Application -Quality of Life | at 6 months
  Efficacy of the smart phone application on patient quality of life will be assessed by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C-30) scores.
Efficacy of Smart Phone Application - Patient Knowledge | Weekly, beginning at baseline to month 6
  Efficacy of the smart phone application on patient knowledge of their diagnosis and treatment will be assessed by weekly true/false quizzes.

CONTACTS AND LOCATIONS:
Overall Officials: Jad Chahoud, MD, MPH, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- [Derived] Roman Souza G, Turner K, Gullapalli K, Paravathaneni M, Ionescu F, Semaan A, DeJesus AB, Trujillo G, Le C, Kim Y, Sun X, Raymond S, Schneider A, Manley B, Jain R, Gilbert S, Jim HSL, Spiess PE, Chahoud J. Feasibility of a Smartphone Application for Education and Symptom Management of Patients With Renal Cell Carcinoma on Combined Tyrosine Kinase and Immune Checkpoint Inhibitors. JCO Clin Cancer Inform. 2024 Jul;8:e2400044. doi: 10.1200/CCI.24.00044. PMID 39058967
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinical-trials-research/clinical-trials/?gclid=EAIaIQobChMImIymzIa-9gIVAZ2GCh3uzAWJEAAYASAAEgI0ovD_BwE